CLINICAL TRIAL: NCT01653730
Title: A Comparative Pilot Study of the Efficacy of Three Portable Oxygen Concentrators During a 6-Minute Walk Test in Patients With Chronic Lung Disease
Brief Title: Comparative Study of 3 Portable Oxygen Concentrators During a 6-minute Walk Test in Patients With Chronic Lung Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Institute for Rehabilitation Research and Development, The Ottawa Hospital Rehabilitation Centre (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: POC-325
Record Dates: First submitted 2012-07-16; First posted 2012-07-31 (Estimated); Last update posted 2012-07-31 (Estimated); Status verified 2012-07

CONDITIONS: Chronic Obstructive Lung Disease; Pulmonary Fibrosis
Keywords: portable oxygen concentrator; 6-minute walk test; chronic obstructive lung disease; pulmonary fibrosis; long term oxygen therapy
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Pulmonary Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Eclipse 3 portable oxygen concentrator (Experimental): Use of the Eclipse 3 portable oxygen concentrator set at maximum pulse-dose setting 10-minutes prior to, and during a 6-minute walk test.
  Interventions: Device: Eclipse 3 portable oxygen concentrator
- iGo portable oxygen concentrator (Experimental): Use of the iGo portable oxygen concentrator set at maximum pulse-dose setting 10-minutes prior to, and during a 6-minute walk test.
  Interventions: Device: iGo portable oxygen concentrator
- EverGo portable oxygen concentrator (Experimental): Use of the iGo portable oxygen concentrator set at maximum pulse-dose setting 10-minutes prior to, and during a 6-minute walk test.
  Interventions: Device: EverGo portable oxygen concentrator
- Control portable oxygen concentrator (No Intervention): 6-minute walk test completed using each patient's own oxygen delivery system set at their usual oxygen prescription for exercise

INTERVENTIONS:
Device: Eclipse 3 portable oxygen concentrator
  Other Names: Eclipse 3 (SeQual Technologies, San Diego, CA, USA)
  Arms: Eclipse 3 portable oxygen concentrator
Device: EverGo portable oxygen concentrator
  Other Names: EverGo (Respironics Inc., Murrysville, PA, USA)
  Arms: EverGo portable oxygen concentrator
Device: iGo portable oxygen concentrator
  Other Names: iGo (DeVillbiss Healthcare, Summerset, PA, USA)
  Arms: iGo portable oxygen concentrator

SUMMARY:
Background: Portable oxygen concentrators (POCs) featuring the latest integrated oxygen conserving devices (OCDs) provide greater patient accessibility and mobility during ambulation and travel. Recent POCs are compact, lightweight, battery-operated, and require no refill-time, thus meeting patients' clinical and lifestyle needs. There is, however, a lack of research on the clinical performance of the latest POCs that could help to determine their ability to maintain patients' oxygen saturations ≥ 90 % during exercise.

Aim: The purpose of this study is to compare the ability of three POCs, with maximum oxygen production capabilities of 950 to 3000 ml per minute, to maintain oxygen saturations ≥ 90 % in patients with chronic lung disease during exercise.

Method: Six minute walk tests (6-MWTs) will be administered in order to measure oxygen saturations by pulse oximetry (SpO2) in up to 20 patients with a diagnosis of either Chronic Obstructive Pulmonary Disease (COPD), or Pulmonary Fibrosis (PF) with documented exertional oxygen desaturations of ≤ 85% on room air. All participants will participate in 4 different 6-minute walk tests: the first will be a control walk performed with the participants' current oxygen system set at their prescribed exertional flow rate. Then, the participants will perform a walk test with each of the three POCs set at the units' maximum pulse dose setting. The order in which the participants use the POCs will be randomly assigned using a sequence generator.

Hypothesis: It is hypothesized that all three POCs will provide oxygen saturations ≥ 90 % during exercise in patients with chronic lung disease with moderate to severe exertional oxygen desaturation.

DETAILED DESCRIPTION:
Participants will attend two study sessions. During the session 1 participants will perform a 6-minute walk test on room air oxygen to assess their suitability for the study. Only those participants with documented exertional oxygen desaturations of ≤ 85% as measured by pulse oximetry during this walk will be asked to return for the second session. During session 2 participants will perform a further four 6-minute walk tests spread over a morning and afternoon testing session. All all data for primary and secondary outcomes will be measured at session 2.

ELIGIBILITY:
Inclusion Criteria:

* Existing diagnosis of chronic obstructive lung disease or pulmonary fibrosis
* completed the pulmonary rehabilitation program at The Ottawa Hospital Rehabilitation Centre between January 30th 2008 and March 31st 2011
* medically stable
* medical prescription for long term oxygen therapy
* 18 years or older

Exclusion Criteria:

* non-ambulatory
* not independent for activities of daily living
* not active in the community
* show limited improvement with any level of continuous oxygen flow rate
* require more than 6 litres per minute of oxygen on continuous flow during exertion
* experienced an exacerbation of their respiratory medical condition over the last 6 weeks, or have not fully recovered from a recent exacerbation
* have moderate to severe orthopaedic or neurological conditions limiting their ability to walk
* have any other impairments that could affect the consistency of the 6-minute walk test
* have severe co-morbid conditions
* are limited by their cardiac condition or have been diagnosed with a cardiac condition since completion of their pulmonary rehabilitation
* severe cognitive or memory deficit
* speak neither French nor English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-02; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Change in saturation of oxygen in the blood after a 6-minute walk test | During study session 2: immediately before beginning (pre-) and immediately after finishing (post-) each of four 6-minute walk tests
  For patient safety oxygen saturation was monitored throughout each 6-minute walk test using pulse oximetry. Pre- and post-walk values were captured as the primary outcome measure.

SECONDARY OUTCOMES:
Total distance walked | During study session 2: immediately after finishing (post-) each of four 6-minute walk tests
Change in Dyspnea ratings after a 6-minute walk test | During study session 2: immediately before beginning (pre-) and immediately after finishing (post-) each of four 6-minute walk tests
  Measured with the modified 10-point Borg scale
Patient preference ratings | During study session 2: immediately after finishing (post-) each of four 6-minute walk tests
  Measured using a self-report questionnaire where patients were asked to indicate how much they agreed with statements about the device they had just used.
Walk time spent with oxygen saturation greater than or equal to 90% | During study session 2: immediately after finishing (post-) each of four 6-minute walk tests

CONTACTS AND LOCATIONS:
Overall Officials: Lyne Lavallée, BSc(PT), Principal Investigator — The Ottawa Hospital Rehabilitation Centre; Carole Leblanc, RRT, Principal Investigator — The Ottawa Hospital Rehabilitation Centre; Doug McKim, MD, Principal Investigator — The Ottawa Hospital
Locations (1):
- The Ottawa Hospital Rehabilitation Centre, Ottawa, Ontario, Canada

REFERENCES:
- [Derived] Leblanc CJ, Lavallee LG, King JA, Taylor-Sussex RE, Woolnough A, McKim DA. A comparative study of 3 portable oxygen concentrators during a 6-minute walk test in patients with chronic lung disease. Respir Care. 2013 Oct;58(10):1598-605. doi: 10.4187/respcare.02275. Epub 2013 Apr 2. PMID 23550171